CLINICAL TRIAL: NCT01302938
Title: Exploratory, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Single Center, Web-Based Phase IV Pilot Methodology Trial To Evaluate The Efficacy And Safety Of Tolterodine ER In Subjects With Overactive Bladder
Brief Title: Web-based Methodology Trial to Evaluate the Efficacy and Safety of Tolterodine ER in Subjects With Overactive Bladder
Acronym: REMOTE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stop date for randomization: 31/5/2012. Recruitment terminated due to lack of recruitment. No new safety issues were identified.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6121195
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Results first posted 2013-09-24 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Overactive Bladder
Keywords: Double-blind; Placebo-controlled; frequency; urgency; web-based; incontinence; methodology; ediary; safety; efficacy; tolerability ER; overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolterodine ER (Experimental)
  Interventions: Drug: Tolterodine ER
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolterodine ER — One 4 mg capsule will be taken with water every day with or without food. It should be swallowed whole without chewing.
  Arms: Tolterodine ER
Drug: Placebo — A placebo of Tolterodine ER 4 mg will be taken with water every day with or without food. It should be swallowed whole without chewing.
  Arms: Placebo

SUMMARY:
To compare the effect of tolterodine ER 4 mg to placebo on patient reported outcomes in subjects with overactive bladder after 1, 4, and 12 weeks of treatment using an innovative web-based trial design

ELIGIBILITY:
Inclusion Criteria:

* Female and 21 years or older
* Overactive bladder symptoms (subject-reported) for at least 3 months
* Be resident in the United States of America and have access and be able to use a computer with internet access throughout the duration of the study

Exclusion Criteria:

* Clinically significant hepatic, renal or neurological condition such as stroke (with residual deficit), multiple sclerosis, spinal cord injury, or Parkinson's disease.
* History of cystitis, continence, urogenitalcancer or radiation
* Subjects who are pregnant, nursing, or with a positive urine pregnancy test or who are intending to become pregnant within 28 days after the completion of the trial.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Mytrus, Inc., San Francisco, California
  - University of California San Francisco, San Francisco, California

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Orri M, Lipset CH, Jacobs BP, Costello AJ, Cummings SR. Web-based trial to evaluate the efficacy and safety of tolterodine ER 4 mg in participants with overactive bladder: REMOTE trial. Contemp Clin Trials. 2014 Jul;38(2):190-7. doi: 10.1016/j.cct.2014.04.009. Epub 2014 May 2. PMID 24792229
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121195&StudyName=Web-based%20Methodology%20Trial%20to%20Evaluate%20the%20Efficacy%20and%20Safety%20of%20Tolterodine%20ER%20in%20Subjects%20with%20Overactive%20Bladder%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 237 participants screened, 118 participants received single-blind placebo matched to tolterodine 4 milligram (mg) capsule once daily during run-in period for 2 weeks. Only 18 participants were randomized to receive double-blind treatment due to early termination of the study.
Groups:
- Tolterodine: Tolterodine 4 mg extended release capsule once daily for 12 weeks.
- Placebo: Placebo matched to tolterodine 4 mg extended release capsule once daily for 12 weeks.
Period: Overall Study
Arm/Group | Tolterodine | Placebo
Started | 12 | 6
Completed | 10 | 6
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolterodine | Placebo | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Customized [Number; unit: participants]
  18 to 44 years | 4 | 3 | 7
  45 to 64 years | 7 | 3 | 10
  Greater than or equal to (>=) 65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 12
Description: Micturitions include episodes of voluntary micturition and episodes of Urgency Urinary Incontinence (UUI). UUI episodes were defined as those micturitions with Urinary Sensation Scale (USS) rating of 5 in the diary in participants with UUI at baseline. USS rating 5: Unable to hold; leak urine. The mean number of micturitions per 24 hours was calculated as the total number of micturitions divided by the total number of diary days collected at that visit.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study medication and had at least 1 baseline or post-baseline efficacy assessment. Missing values imputed using Last observation carried forward (LOCF) method. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 11 | 6
micturitions per 24 hours
  Baseline | 11.5 (3.5) | 9.9 (1.7)
  Change at Week 12 | -2.6 (2.3) | -0.3 (2.3)
Statistical Analysis 1: Comparison: Tolterodine vs Placebo; Change at Week 12: Analysis was performed using an analysis of covariance (ANCOVA) with term for treatment with baseline value as a covariate; Test type: Superiority or Other; Least squares (LS) mean difference = -1.6, 95% CI 2-sided [-3.9 to 0.6], Standard Error of Mean 1.0

2. Secondary Outcome: Change From Baseline in Mean Voided Volume Per Micturition at Week 1, 4 and 12
Description: Mean voided volume per micturition was calculated as sum of voided volume divided by the total number of micturition episodes with a recorded voided volume greater than 0 at that visit. Baseline values for each time point were calculated separately considering only those participants who were evaluable at the given time point.
Time Frame: Baseline, Week 1, 4, 12
Population: FAS population. Missing values imputed using LOCF method. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure. 'n' = number of participants who were evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 11 | 6
milliliter (mL)
  Baseline for Week 1 (n=10,5) | 163.7 (59.8) | 194.2 (60.3)
  Baseline for Week 4 (n=11,6) | 161.2 (57.4) | 185.2 (58.3)
  Baseline for Week 12 (n=11,6) | 161.2 (57.4) | 185.2 (58.3)
  Change at Week 1 (n=10,5) | 49.8 (66.3) | 27.9 (51.1)
  Change at Week 4 (n=11,6) | 45.2 (84.0) | 19.2 (41.2)
  Change at Week 12 (n=11,6) | 31.9 (68.3) | -10.1 (30.4)
Statistical Analysis 1: Comparison: Tolterodine vs Placebo; Change at Week 1: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = 29.4, 95% CI 2-sided [-47.8 to 106.6], Standard Error of Mean 35.4
Statistical Analysis 2: Comparison: Tolterodine vs Placebo; Change at Week 4: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = 28.0, 95% CI 2-sided [-55.4 to 111.4], Standard Error of Mean 38.9
Statistical Analysis 3: Comparison: Tolterodine vs Placebo; Change at Week 12: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = 43.0, 95% CI 2-sided [-24.2 to 110.3], Standard Error of Mean 31.4

3. Secondary Outcome: Change From Baseline in Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 1, 4 and 12
Description: UUI episodes were defined as those with the Urinary Sensation Scale (USS) rating of 5 in the diary. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. Baseline values for each time point were calculated separately considering only those participants who were evaluable at the given time point.
Time Frame: Baseline, Week 1, 4, 12
Population: as for outcome 2
Measure: Median (Full Range); unit: episodes per 24 hours
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 11 | 6
episodes per 24 hours
  Baseline for Week 1 (n=10,5) | 3.2 [1.0 to 7.7] | 2.3 [1.0 to 5.7]
  Baseline for Week 4 (n=11,6) | 2.7 [1.0 to 7.7] | 2.3 [1.0 to 5.7]
  Baseline for Week 12 (n=11,6) | 2.7 [1.0 to 7.7] | 2.3 [1.0 to 5.7]
  Change at Week 1 (n=10,5) | -1.0 [-2.3 to 1.7] | -0.7 [-2.7 to -0.3]
  Change at Week 4 (n=11,6) | -1.3 [-5.3 to 0.3] | -1.9 [-3.7 to -0.7]
  Change at Week 12 (n=11,6) | -1.7 [-7.7 to 0.0] | -1.2 [-3.0 to 0.3]
Statistical Analysis 1: Comparison: Tolterodine vs Placebo; Change at Week 1: Non-parametric Hodges-Lehmann's method was used to obtain median difference and 95 percent (%) confidence intervals (CI); Test type: Superiority or Other; Median Difference (Final Values) = 0.17, 95% CI 2-sided [-0.67 to 1.67]
Statistical Analysis 2: Comparison: Tolterodine vs Placebo; Change at Week 4: Non-parametric Hodges-Lehmann's method was used to obtain median difference and 95% CI; Test type: Superiority or Other; Median Difference (Final Values) = 0.58, 95% CI 2-sided [-1.00 to 1.83]
Statistical Analysis 3: Comparison: Tolterodine vs Placebo; Change at Week 12: Non-parametric Hodges-Lehmann's method was used to obtain median difference and 95% CI; Test type: Superiority or Other; Median Difference (Final Values) = -0.50, 95% CI 2-sided [-3.00 to 1.00]

4. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 1 and 4
Description: Micturitions include episodes of voluntary micturition and episodes of UUI. UUI episodes were defined as those micturitions with USS rating of 5 in the diary in participants with UUI at baseline. USS rating 5: Unable to hold; leak urine. The mean number of micturitions per 24 hours was calculated as the total number of micturitions divided by the total number of diary days collected at that visit. Baseline values for each time point were calculated separately considering only those participants who were evaluable at the given time point.
Time Frame: Baseline, Week 1, 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 11 | 6
micturitions per 24 hours
  Baseline for Week 1 (n=10,5) | 11.7 (3.6) | 9.9 (1.8)
  Baseline for Week 4 (n=11,6) | 11.5 (3.5) | 9.9 (1.7)
  Change at Week 1 (n=10,5) | -0.6 (1.2) | -0.7 (1.4)
  Change at Week 4 (n=11,6) | -2.4 (2.2) | -1.0 (0.9)
Statistical Analysis 1: Comparison: Tolterodine vs Placebo; Change at Week 1: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = 0.3, 95% CI 2-sided [-1.3 to 1.8], Standard Error of Mean 0.7
Statistical Analysis 2: Comparison: Tolterodine vs Placebo; Change at Week 4: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = -0.6, 95% CI 2-sided [-2.2 to 0.9], Standard Error of Mean 0.7

5. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Micturitions Per 24 Hours at Week 1, 4 and 12
Description: Nocturnal micturitions were defined as micturitions with USS rating 1-5 that occurred between the time the participant went to bed and the time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. The mean number of nocturnal micturitions per 24 hours was calculated as the total number of nocturnal micturitions divided by the total number of diary days collected at that visit.
Time Frame: Baseline, Week 1, 4, 12
Population: Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis, as per change in planned analysis.
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Micturition-Related Urgency Episodes Per 24 Hours at Week 1, 4 and 12
Description: The mean number of micturition-related nocturnal urgency episodes per 24 hours was calculated as the total number of micturitions with USS rating of greater than or equal to (>=) 3 that occurred between time participant went to bed and time participant arose to start next day divided by the total number of days that diary data was collected at that visit. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Week 1, 4, 12
Population: as for outcome 5
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Mean Number of Micturition-Related Urgency Episodes Per 24 Hours at Week 1, 4 and 12
Description: The mean number of micturition-related urgency episodes per 24 hours was calculated as the total number of micturitions with USS rating of >= 3 divided by the total number of days that diary data was collected at that visit. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. Baseline values for each time point were calculated separately considering only those participants who were evaluable at the given time point.
Time Frame: Baseline, Week 1, 4, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 11 | 6
episodes per 24 hours
  Baseline for Week 1 (n=10,5) | 9.1 (2.2) | 8.5 (3.1)
  Baseline for Week 4 (n=11,6) | 9.0 (2.1) | 8.1 (3.0)
  Baseline for Week 12 (n=11,6) | 9.0 (2.1) | 8.1 (3.0)
  Change at Week 1 (n=10,5) | -1.1 (1.2) | -1.6 (0.8)
  Change at Week 4 (n=11,6) | -3.2 (2.1) | -1.6 (1.9)
  Change at Week 12 (n=11,6) | -3.9 (2.8) | -1.0 (3.1)
Statistical Analysis 1: Comparison: Tolterodine vs Placebo; Change at Week 1: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = 0.6, 95% CI 2-sided [-0.8 to 1.9], Standard Error of Mean 0.6
Statistical Analysis 2: Comparison: Tolterodine vs Placebo; Change at Week 4: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = -1.4, 95% CI 2-sided [-3.7 to 0.8], Standard Error of Mean 1.1
Statistical Analysis 3: Comparison: Tolterodine vs Placebo; Change at Week 12: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = -2.9, 95% CI 2-sided [-6.3 to 0.4], Standard Error of Mean 1.5

8. Secondary Outcome: Number of Participants With Change From Baseline in Patient Perception of Bladder Condition (PPBC) at Week 1, 4 and 12
Description: PPBC: self-administered,single-item questionnaire to describe participant's perception of bladder-related problems. PPBC assessed on 6-point scale:1=no problems at all,2=some very minor problems,3=some minor problems,4=some moderate problems,5=severe problems,6=many severe problems. Results categorized as score change (SC) from baseline on 2-point scale:improvement (negative SC),no improvement (SC 0 or more) and on 4-point scale:major improvement (SC is negative in magnitude of 2 or more), minor improvement (SC is negative in magnitude of 1), no change (SC= 0),deterioration (positive SC).
Time Frame: Baseline, Week 1, 4, 12
Population: FAS included all participants who received at least 1 dose of study medication and had at least 1 baseline or post-baseline efficacy assessment. Missing values imputed using LOCF method. 'n' = number of participants who were evaluable at specific time points for each arm group, respectively.
Measure: Number; unit: participants
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 12 | 6
participants
  Baseline, Week 1: No Problems at all (n=11,5) | 0 | 0
  Baseline, Week 1:Some Very Minor Problems(n=11,5) | 0 | 0
  Baseline, Week 1: Some Minor Problems (n=11,5) | 1 | 1
  Baseline, Week 1:Some Moderate Problems(n=11,5) | 2 | 2
  Baseline, Week 1: Severe Problems (n=11,5) | 8 | 1
  Baseline, Week 1: Many Severe Problems (n=11,5) | 0 | 1
  Baseline, Week 4: No Problems at all (n=12,6) | 0 | 0
  Baseline, Week 4: Some Very Minor Problems(n=12,6) | 0 | 0
  Baseline, Week 4: Some Minor Problems (n=12,6) | 1 | 2
  Baseline, Week 4: Some Moderate Problems (n=12,6) | 3 | 2
  Baseline, Week 4: Severe Problems (n=12,6) | 8 | 1
  Baseline, Week 4: Many Severe Problems (n=12,6) | 0 | 1
  Baseline, Week 12: No Problems at all (n=12,6) | 0 | 0
  Baseline, Week12: Some Very Minor Problems(n=12,6) | 0 | 0
  Baseline, Week 12: Some Minor Problems (n=12,6) | 1 | 2
  Baseline, Week 12: Some Moderate Problems (n=12,6) | 3 | 2
  Baseline, Week 12: Severe Problems (n=12,6) | 8 | 1
  Baseline, Week 12: Many Severe Problems (n=12,6) | 0 | 1
  Week 1:Improvement (2-point scale) (n=11,5) | 7 | 2
  Week 1:No improvement (2-point scale) (n=11,5) | 4 | 3
  Week 1:Major improvement (4-point scale) (n=11,5) | 2 | 1
  Week 1:Minor improvement (4-point scale) (n=11,5) | 5 | 1
  Week 1:No Change (4-point scale) (n=11,5) | 3 | 1
  Week 1:Deterioration (4-point scale) (n=11,5) | 1 | 2
  Week 4:Improvement (2-point scale) (n=12,6) | 7 | 3
  Week 4:No improvement (2-point scale) (n=12,6) | 5 | 3
  Week 4:Major improvement (4-point scale) (n=12,6) | 4 | 1
  Week 4:Minor improvement (4-point scale) (n=12,6) | 3 | 2
  Week 4:No Change (4-point scale) (n=12,6) | 5 | 2
  Week 4:Deterioration (4-point scale) (n=12,6) | 0 | 1
  Week 12:Improvement (2-point scale) (n=12,6) | 9 | 4
  Week 12:No improvement (2-point scale) (n=12,6) | 3 | 2
  Week 12:Major improvement (4-point scale) (n=12,6) | 7 | 1
  Week 12:Minor improvement (4-point scale) (n=12,6) | 2 | 3
  Week 12:No Change (4-point scale) (n=12,6) | 3 | 2
  Week 12:Deterioration (4-point scale) (n=12,6) | 0 | 0

9. Secondary Outcome: Number of Participants With Change From Baseline in Patient Perception of Urgency Scale (PPUS) at Week 1, 4 and 12
Description: PPUS: a self-administered, single-item, validated questionnaire that measures the participant's perception of urinary urgency. It is sensitive to changes in perceptions of urinary urgency over time. Scale of 0 (usually not able to hold urine), 1 (usually able to hold urine [without leaking] until reaching toilet if go to toilet immediately), or 2 (usually able to finish what he/she is doing before going to toilet [without leaking]). Results categorized as SC from baseline on 3-point scale: improvement (positive SC), no change (SC 0), deterioration (negative SC).
Time Frame: Baseline (Bl), Week 1, 4, 12
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 12 | 6
participants
  Bl,Week 1:Not able to hold urine (n=11,5) | 6 | 1
  Bl,Week 1:Able to hold until reach toilet (n=11,5) | 4 | 3
  Bl,Week 1:Able to finish what I am doing (n=11,5) | 1 | 1
  Bl,Week 4:Not able to hold urine (n=12,6) | 6 | 1
  Bl,Week 4:Able to hold until reach toilet (n=12,6) | 5 | 4
  Bl,Week 4:Able to finish what I am doing (n=12,6) | 1 | 1
  Bl,Week 12:Not able to hold urine (n=12,6) | 6 | 1
  Bl,Week 12:Able to hold until reach toilet(n=12,6) | 5 | 4
  Bl,Week 12:Able to finish what I am doing (n=12,6) | 1 | 1
  Week 1:Improvement (n=11,5) | 4 | 1
  Week 1:No change (n=11,5) | 6 | 3
  Week 1:Deterioration (n=11,5) | 1 | 1
  Week 4:Improvement (n=12,6) | 4 | 0
  Week 4:No change (n=12,6) | 7 | 5
  Week 4:Deterioration (n=12,6) | 1 | 1
  Week 12:Improvement (n=12,6) | 6 | 1
  Week 12:No change (n=12,6) | 6 | 4
  Week 12:Deterioration (n=12,6) | 0 | 1

10. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score at Week 12
Description: OAB-q: a self-administered, 33-item, questionnaire that assesses how much the participant has been bothered by selected bladder symptoms. Each item rated by participant on Likert scale 1 (not at all) to 6 (a very great deal). Symptom bother score derived as sum of scores for items 1 to 8; lowest possible raw score: 8; highest possible score: 48. Data analyzed based on transformation of the score to a 0 to 100 scale [(Actual total raw score - lowest possible value of raw score)/range]*100. Higher scores values indicative of greater symptom bother.
Time Frame: Baseline, Week 12
Population: FAS included all participants who received at least 1 dose of study medication and had at least 1 baseline or post-baseline efficacy assessment. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 10 | 6
units on a scale
  Baseline | 66.5 (25.8) | 54.6 (32.7)
  Change at Week 12 | -27.8 (21.8) | -12.5 (25.8)
Statistical Analysis 1: Comparison: Tolterodine vs Placebo; Change at Week 12: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = -10.0, 95% CI 2-sided [-33.2 to 13.2], Standard Error of Mean 10.8

11. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL) Domains and Total Score of Overactive Bladder Questionnaire (OAB-q) at Week 12
Description: OAB-q: self-administered, 33-item, questionnaire, assesses how much participant has been bothered by selected bladder symptoms. Each item rated on Likert scale 1 (not at all) to 6 (a very great deal). Questions 9 to 33 constitute HRQL, includes domains (range): concern(7-42), coping(8-48), sleep(5-30), and social function(5-30). Total HRQL score (25-125) derived as sum of HRQL domains. Transformed score range 0 to 100 (HRQL domain or total) = [(Highest possible raw score-Actual total raw score)/Raw score range]*100. Higher transformed scores indicate better HRQL.
Time Frame: Baseline, Week 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 10 | 6
units on a scale
  Baseline: Coping Subscale | 50.0 (25.9) | 56.3 (33.3)
  Baseline: Concern Subscale | 41.7 (25.8) | 53.8 (37.2)
  Baseline: Sleep Subscale | 49.2 (32.2) | 55.3 (38.0)
  Baseline: Total HRQL Score | 54.1 (21.1) | 58.5 (35.1)
  Change at Week 12: Coping Subscale | 26.3 (19.0) | 13.8 (10.1)
  Change at Week 12: Concern Subscale | 29.4 (25.8) | 16.7 (20.8)
  Change at Week 12: Sleep Subscale | 21.6 (31.2) | 8.0 (19.4)
  Change at Week 12: Total HRQL Score | 22.5 (21.6) | 12.0 (14.4)
Statistical Analysis 1: Comparison: Tolterodine vs Placebo; Change at Week 12; Coping Subscale: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = 11.7, 95% CI 2-sided [-6.9 to 30.3], Standard Error of Mean 8.6
Statistical Analysis 2: Comparison: Tolterodine vs Placebo; Change at Week 12; Concern Subscale: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = 8.0, 95% CI 2-sided [-16.7 to 32.7], Standard Error of Mean 11.4
Statistical Analysis 3: Comparison: Tolterodine vs Placebo; Change at Week 12; Sleep Subscale: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = 10.3, 95% CI 2-sided [-13.3 to 33.8], Standard Error of Mean 10.9
Statistical Analysis 4: Comparison: Tolterodine vs Placebo; Change at Week 12; Total HRQL Score: Analysis was performed using an ANCOVA with term for treatment with baseline value as a covariate; Test type: Superiority or Other; LS mean difference = 9.0, 95% CI 2-sided [-11.0 to 29.0], Standard Error of Mean 9.3

12. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL) Social Domain Score at Week 12
Description: as for outcome 11
Time Frame: Baseline, Week 12
Population: as for outcome 10
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 10 | 6
units on a scale
  Baseline | 84.0 [56.0 to 100.0] | 92.0 [20.0 to 100.0]
  Change at Week 12 | 10.0 [-32.0 to 36.0] | 2.0 [-4.0 to 36.0]
Statistical Analysis 1: Comparison: Tolterodine vs Placebo; Change at Week 12; Social Subscale: Non-parametric Hodges-Lehmann's method was used to obtain median difference and 95% CI; Test type: Superiority or Other; Median Difference (Final Values) = 4.00, 95% CI 2-sided [-20.00 to 20.00]

13. Secondary Outcome: Number of Participants With Response Regarding Source of First Information About Study
Description: Participant experience questionnaire (PEQ) is a web-based self-administered, exploratory questionnaire that assesses the participant's perception of trial method. Number of participants who responded to question 1, "Where did you hear first about the study?" are reported.
Time Frame: Week 12
Population: FAS included all participants who received at least 1 dose of study medication and had at least 1 baseline or post-baseline efficacy assessment. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: participants
Groups:
- Entire Study Population: Includes all participants who received either tolterodine 4 mg extended release capsule once daily or matching placebo for 12 weeks.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 17
participants
  Friend | 2
  Google or related internet search engine | 3
  Web-site advertisement | 3
  Blogger, on-line health group leader or activist | 1
  On-line Community | 1
  Email | 3
  Other | 4

14. Secondary Outcome: Number of Participants With Reason for Participation in the Study
Description: PEQ is a web-based self-administered, exploratory questionnaire that assesses the participant's perception of trial method. Number of participants who responded to question 2, "What led you to participate given the study drug is already available?" are reported.
Time Frame: Week 12
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 17
participants
  Contribute to research | 8
  Experience internet research study and try it out | 2
  Ease of participation | 3
  Free medication | 3
  Payment for participation | 1

15. Secondary Outcome: Participant Perception Regarding Satisfaction Related to Study
Description: PEQ:self-administered, to assess perception of trial method. Question3, "How satisfied were you with items?" on scale 1(very satisfied) to 5(very dissatisfied)- recruitment; questionnaires,surveys(Ques,Sur); identification verification(IV); informed consent(IC) process; website experience; phone call; laboratory(lab) kit delivery; lab location; lab staff service(Ser); physical exam(PE) scheduling,location (sch,loc); PE visit; medication(med) first batch delivery; med second batch delivery; cell phone(CP) received; CP use; call center(CC) ser; medical support(supp); technical supp; overall.
Time Frame: Week 12
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 17
participants
  Recruitment: neither dis-satisfied nor satisfied | 1
  Recruitment: somewhat satisfied | 4
  Recruitment: very satisfied | 12
  Ques,Sur: somewhat dis-satisfied | 1
  Ques,Sur: somewhat satisfied | 4
  Ques,Sur: very satisfied | 12
  IV: somewhat dis-satisfied | 1
  IV: neither dis-satisfied nor satisfied | 2
  IV: somewhat satisfied | 3
  IV: very satisfied | 11
  IC: somewhat dis-satisfied | 1
  IC: neither dis-satisfied nor satisfied | 1
  IC: somewhat satisfied | 2
  IC: very satisfied | 13
  Website experience: very dis-satisfied | 2
  Website experience: somewhat satisfied | 4
  Website experience: very satisfied | 11
  Phone call: very dis-satisfied | 1
  Phone call: somewhat dis-satisfied | 1
  Phone call: somewhat satisfied | 1
  Phone call: very satisfied | 14
  Lab kit delivery: very dis-satisfied | 1
  Lab kit delivery: very satisfied | 16
  Lab location: neither dis-satisfied nor satisfied | 3
  Lab location: somewhat satisfied | 1
  Lab location: very satisfied | 13
  Lab staff Ser: neither dis-satisfied nor satisfied | 1
  Lab staff Ser: somewhat satisfied | 3
  Lab staff Ser: very satisfied | 13
  PE sch,loc: somewhat dis-satisfied | 2
  PE sch,loc: neither dis-satisfied nor satisfied | 3
  PE sch,loc: very satisfied | 12
  PE visit: very dis-satisfied | 1
  PE visit: somewhat dis-satisfied | 2
  PE visit: neither dis-satisfied nor satisfied | 2
  PE visit: somewhat satisfied | 1
  PE visit: very satisfied | 11
  Med first batch delivery: very dis-satisfied | 1
  Med first batch delivery: very satisfied | 16
  Med second batch delivery: very dis-satisfied | 1
  Med second batch delivery: somewhat satisfied | 1
  Med second batch delivery: very satisfied | 15
  CP received: very satisfied | 17
  CP use: very dis-satisfied | 1
  CP use: neither dis-satisfied nor satisfied | 1
  CP use: somewhat satisfied | 1
  CP use: very satisfied | 14
  CC ser: neither dis-satisfied nor satisfied | 4
  CC ser: somewhat satisfied | 1
  CC ser: very satisfied | 12
  Medical supp: somewhat dis-satisfied | 1
  Medical supp: somewhat satisfied | 1
  Medical supp: very satisfied | 15
  Technical supp:neither dis-satisfied nor satisfied | 2
  Technical supp: somewhat satisfied | 1
  Technical supp: very satisfied | 14
  Overall: somewhat dis-satisfied | 2
  Overall: somewhat satisfied | 4
  Overall: very satisfied | 11

16. Secondary Outcome: Participant Perception Regarding Cell Phone Diary
Description: PEQ:self-administered, assesses participants perception of trial method. Question4, "How satisfied were you with items?" on scale 1(very easy) to 5(very difficult)- a: teaching video explaining CP use; recording urinations using CP; size of text on CP; sending your urinary information(inf) using your CP, e: overall, suitability for capturing urinations as they happened.
Time Frame: Week 12
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 17
participants
  CP use video: neither difficult nor easy | 1
  CP use video: somewhat easy | 4
  CP use video: very easy | 12
  Recording urinations using CP: somewhat easy | 3
  Recording urinations using CP: very easy | 14
  CP text size: neither difficult nor easy | 1
  CP text size: somewhat easy | 4
  CP text size: very easy | 12
  Sending urinary inf using CP: somewhat easy | 4
  Sending urinary inf using CP: very easy | 13
  Overall: neither difficult nor easy | 1
  Overall: somewhat easy | 3
  Overall: very easy | 13

17. Secondary Outcome: Participant Perception Regarding Received Treatment in the Study
Description: PEQ is a web-based self-administered, exploratory questionnaire that assesses the participant's perception of trial method. Number of participants who responded to question 5, "What treatment did you think you were on?" are reported.
Time Frame: Week 12
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 11 | 6
participants
  Placebo | 3 | 4
  Tolterodine | 8 | 2

18. Secondary Outcome: Participant Perception Regarding Recommending a Friend to Enter Similar Study
Description: PEQ is a web-based self-administered, exploratory questionnaire that assesses the participant's perception of trial method. Number of participants who responded to question 6, "How likely would you be to recommend a friend to enter a similar study?" are reported.
Time Frame: Week 12
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 17
participants
  Very likely | 11
  Somewhat likely | 5
  Neither | 1

19. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 28 days after last dose
Population: Safety set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 12 | 6
participants
  AEs | 6 | 3
  SAEs | 0 | 0

20. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) by Relatedness and Severity
Description: AE:any untoward medical occurrence attributed to study medication in participant who received study drug. Relatedness to study medication was assessed by the investigator. Severity of AEs assessed as: mild (does not interfere with participant's usual function), moderate (interferes to some extent with participant's usual function) and severe (interferes significantly with participant's usual function). Mild, moderate and severe are not mutually exclusive; hence same participant may be included in more than 1 type of severity of AEs.
Time Frame: Baseline up to 28 days after last dose
Population: Safety set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 12 | 6
participants
  Treatment-related AEs | 2 | 0
  Mild AEs | 4 | 3
  Moderate AEs | 3 | 0
  Severe AEs | 1 | 0

21. Other Pre Specified Outcome: Number of Participants Who Discontinued the Study Due to Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to 28 days after last dose
Population: Safety set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 12 | 6
participants | 1 | 0

22. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria for potentially clinically significant (PCS) laboratory values: Hemoglobin, hematocrit, red blood cell less than (<) 0.8 lower limit of normal(LLN); platelet <0.5 LLN, >1.75 upper LN (ULN);white blood cell <0.6 LLN, >1.5 ULN; lymphocyte, total neutrophil(absolute[AL]),Total protein, albumin, phosphate <0.8 LLN, >1.2 ULN; basophil, eosinophil, monocyte >1.2ULN; Total bilirubin >1.5ULN; aspartate, alanine aminotransferase, alkaline phosphatase >3ULN; Blood urea nitrogen, creatinine >1.3ULN; sodium <0.95LLN, >1.05ULN; potassium, chloride, bicarbonate, calcium <0.9LLN, >1.1ULN.
Time Frame: Week 12
Population: Safety set included all participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 10 | 6
participants | 1 | 1

ADVERSE EVENTS:
Arm/Group | Tolterodine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 1/12 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolterodine (N=12) | Placebo (N=6)
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to low participant enrollment and due to relatively small sample size; results should be interpreted with caution. Early termination of the study was not related to any safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.